CLINICAL TRIAL: NCT07299994
Title: Efficacy and Safety of Intravenous Thrombolysis in Branch Atheromatous Disease - a Retrospective Data Analysis
Brief Title: Efficacy and Safety of Intravenous Thrombolysis in Branch Atheromatous Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Sponsor
Other Study IDs: 17823177
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Thrombolysis; DAPT(Dual Antiplatelet Therapy); SAPT(Single Antiplatelet Therapy); Acute Ischemic Stroke
Keywords: Acute ischemic Stroke; Branch Atheromatous Disease; Thrombolysis; DAPT; SAPT
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IVT group: Patients who received intravenous thrombolysis as part of acute stroke treatment, if eligible.
- Antiplatelet group: Patients who received SAPT or DAPT as part of acute stroke treatment.

SUMMARY:
Rationale and Relevance:

Branch Atheromatous Disease (BAD) describes an atherosclerotic occlusion of one of the deep penetrating cerebral arteries, including the lenticulostriate artery (LSA), paramedian pontine artery (PPA), and anterior choroidal artery (ACHA). BAD is frequently associated with early neurological deterioration (END), particularly progressive motor deficits that contribute to increased disability. Despite its clinical relevance, BAD remains underrepresented in major radiomorphological classification systems such as TOAST, which has led to limited evidence and unclear treatment strategies. Previous studies suggest that the efficacy of intravenous thrombolysis (IVT) may be reduced in BAD compared to other stroke etiologies.

Objectives:

The primary objective of this study is to evaluate the efficacy and safety of IVT compared with single antiplatelet therapy (SAPT) and dual antiplatelet therapy (DAPT) in patients with BAD-related stroke. A secondary objective is to examine the impact of acute-phase blood pressure fluctuations on END and functional neurological outcomes.

Design and Methods:

This international multicenter study will be conducted retrospectively according to the STROBE guidelines. Eligible patients include those with BAD-related stroke treated at one of the participating centers between 2010 and 2025. Inclusion criteria comprise characteristic diffusion-weighted MRI patterns in predefined vascular territories (LSA, PPA, ACHA) and a symptom onset ≤24 hours before admission. Patients with typical lacunar infarcts or with other identified stroke etiologies will be excluded.

Endpoints:

Primary endpoints include functional outcome at three months, defined as a favorable outcome with a modified Rankin Scale score of 0-1; occurrence of END, defined as a ≥4-point worsening on the NIHSS within 24-48 hours; and symptomatic intracerebral hemorrhage. Collected data include clinical, imaging, and therapeutic variables, as well as blood pressure trajectories and pre-stroke treatments (as detailed in the study protocol).

Statistical Analysis:

Analyses will be performed using SPSS and R. Descriptive statistics, univariate analyses, and multivariable models (IPTW and Poisson regression) will be applied. Results will be reported as adjusted relative risks with 95% confidence intervals.

Significance:

This study will provide the first comprehensive evaluation of IVT versus SAPT/DAPT in BAD-related stroke, and will investigate the clinical impact of blood pressure changes in this specific stroke subtype. The findings aim to support evidence-based treatment recommendations for a currently underrecognized and poorly understood stroke etiology.

DETAILED DESCRIPTION:
Background Intracranial branch atheromatous disease (BAD) describes an occlusion of deep penetrating intracranial arteries, leading to subcortical infarction. Perforating arteries include the lenticulostriate artery (LSA), paramedian pontine artery (PPA), anterior choroidal artery (ACHA), thalamoperforating artery, and Heubner's artery. This study focuses on BAD affecting the ACHA, LSA, and PPA.

In contrast to lacunar ischemia, which is caused by hypertensive lipohyalinotic degeneration of the distal segment of a perforating artery with a diameter ≤200 µm, BAD involves larger vessels (700-800 µm) affected by atherosclerosis of the parent artery. BAD has not been classified as a major cause of cerebral infarction by the National Institute of Neurological Disorders and Stroke (NINDS) or the Trial of Org 10172 in Acute Stroke Treatment (TOAST), which has contributed to a rather scarce data regarding clinical trajectories of this particular stroke etiology. According to TOAST criteria, BAD-related strokes are often categorized under small vessel occlusion or classified as an undetermined cause. Due to their vessel size, high pressure and flow, these arteries are more susceptible to endothelial damage and atherosclerosis, leading to fluctuating symptoms. At admission, BAD often presents similarly to lacunar ischemia. But in comparison, a main clinical characteristic of BAD is the frequent occurrence of early neurological deterioration (END), often manifesting as progressive motor deficits, which contribute to poorer outcomes and increased disability. Consequently, BAD has been recognized as a major vascular mechanism of progressive motor deficits in penetrating artery infarcts. Because of its unique pathophysiology and clinical progression, finding effective treatment strategies remains difficult. Intravenous thrombolysis (IVT) appears to be less effective for BAD compared to other etiologies of acute ischemic stroke. Previous studies have explored various treatment strategies, including dual antiplatelet therapy, tirofiban, and anticoagulation therapy, but results have been inconsistent. This study will assess the efficacy and safety of IVT versus antiplatelet therapy in BAD-related stroke. Furthermore, we will examine the impact of blood pressure on END and functional outcomes.

Aims The primary aim of this study is to assess the efficacy and safety of IVT compared to single (SAPT) or dual antiplatelet therapy (DAPT) in patients with BAD-related stroke. Secondary aim is to explore the impact of blood pressure fluctuations on END and functional outcomes and its potential interactions with acute therapies.

Methods This study is an international multicenter observational study recruiting patients with BAD-related stroke in the acute phase on the stroke unit up to 24 hours before admission. As of March 26, 2025, this study has recruited six institutions, led by Department of Neurology, St. John's Hospital, Vienna, Austria and sponsored by Sigmund Freud University Vienna, Austria.

Study Population All patients with a BAD-related stroke, aged over 18 years, with symptom onset no more than 24 hours before admission, who were treated in one of the stroke units of the participating institutions between 01.01.2010 and 28.02.2025, will be included based on the following inclusion criteria. All enrolled patients must have undergone a cerebral MRI for inclusion.

Inclusion criteria

1. DWI lesion: single isolated deep subcortical stroke AND
2. The affected vessel involves the LSA, PPA, or ACHA, and the infarct lesion on DWI conforms to one of the following characteristics (A, B, OR C):

A. LSA: "Comma-like" infarct lesions with "fan-shaped" extension from bottom to top in the coronary position OR ≥ 3 layers (layer thickness 5 mm) on axial DWI.

B. PPA: Infarct lesion extending from the deep pons to the ventral pons on axial DWI.

C. ACHA: Infarct within the anterior choroidal artery territory. Exclusion criteria

1. Typical recent small subcortical infarction (RSSI) (oval, <20mm in all axes).
2. ≥ 50% stenosis on the parent artery (i.e., BA, MCA, or ICA)
3. Stroke due to other clearly identified causes or possible cardioembolic etiology.

Endpoints

The primary endpoints of this study include:

1. Modified Rankin Scale (mRS) score at three months, with a favorable outcome defined as mRS 0-1 at three months.
2. Early neurological deterioration (END), defined as a worsening of the NIHSS score by ≥4 points within 24-48 hours after symptom onset.
3. Occurrence of symptomatic intracerebral hemorrhage.

Interventions Intravenous thrombolysis (IVT), single antiplatelet therapy (SAPT), dual antiplatelet therapy (DAPT)

Hypothesis

1. H0. Patients with BAD related stroke treated using IVT will not achieve better functional outcome as compared to those treated with SAPT.

   H1. Patients with BAD related stroke treated using IVT will achieve better functional outcome as compared to those treated with SAPT.
2. H0. Patients with BAD related stroke treated using IVT will not achieve better functional outcome as compared to those treated with DAPT.

   H1. Patients with BAD related stroke treated using IVT will achieve better functional outcome as compared to those treated with DAPT.
3. H3. Patients with BAD-related stroke experiencing blood pressure drop >=30 mmHg in the first 24 hours after admission will not experience worse functional outcome as compared to those without blood pressure drop. Interaction with IVT will be significant.

H3. Patients with BAD-related stroke experiencing blood pressure drop >=30 mmHg in the first 24 hours after admission will experience worse functional outcome as compared to those without blood pressure drop. Interaction with IVT will be significant.

Informed consent Due to the retrospective nature of the study and the use of anonymized data, obtaining patient informed consent is not necessary.

Study sites Institutions participating in this study, with a full list of institutions provided under collaborating institutions. The leading institution is the Department of Neurology, St. John's Hospital, Vienna, Austria.

Study design The study will be conducted as an international multicenter retrospective observational study according to the STROBE guideline.

Sample size Although the study is retrospective, a sample size calculation was conducted. Based on outcome data from lacunar stroke patients, 59% of patients treated with IVT achieved a favorable outcome (mRS 0 - 1 at 3 months). Assuming an odds ratio (OR) of 1.67 in favor of IVT, this corresponds to an estimated 46% rate of favorable functional outcome in the control group. Using a two-sided alpha of 0.05 and a power of 80%, the calculated total sample size is 462 patients, with 231 in each group. The calculation was performed using G*Power (version 3.1.9.7, Düsseldorf, Germany).

Collected data See study protocol

Data management Collected data will be entered into an electronic database at the primary study site. All data will be fully anonymized and only shared in this form with researchers. Therefore, a data monitoring committee will not be required. All datasets will be exclusively used for this study, and no third party will be granted access at any time.

Statistics The statistical analysis will be conducted using SPSS version 29.0.1.0 (IBM Corp., Armonk, NY, USA) and R version 4.4.2 (R Foundation for Statistical Computing, Vienna, Austria). Continuous variables will be presented as mean ± standard deviation (SD) or median with interquartile range (IQR), depending on their distribution. Categorical variables will be expressed as frequencies (n) and percentages (%). This includes variables such as baseline characteristics, medical history, and treatment modalities. For the analysis of statistical significance in outcome measures, Pearson's χ² test or Fisher's exact test will be applied for categorical data, while Wilcoxon rank-sum tests or t-tests will be used for continuous variables, as appropriate. Statistical uncertainty will be reported using 95% confidence intervals (CI). To evaluate the association between three-month mRS and clinical or therapeutic predictors, IPTW and Poisson regression models will be utilized. The results of the Poisson regression analysis will be reported as adjusted relative risks (RR) with corresponding 95% CI. A favorable functional outcome is defined as mRS ≤1 at three months post-stroke. Statistical significance will be set at p<0.05.

Ethical considerations This study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines throughout the whole research process. Approval from the ethics committee will be obtained prior to data collection. As this is a retrospective, non-interventional study, there is no additional physical risk for patients. Data collection is exclusively based on previously recorded medical records. The primary ethical concern in this study relates to data transfer between institutions. To minimize this risk, only fully anonymized data will be shared with researchers. All collected data will be used solely for scientific research purposes, and no personal information will be disclosed or made accessible to third parties.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years, with acute ischemic stroke and symptom onset no more than 24 hours before admission, who were treated in one of the stroke units of the participating institutions.
* All enrolled patients must have undergone a cerebral MRI for inclusion:

  1. DWI lesion: single isolated deep subcortical stroke AND
  2. The affected vessel involves the LSA, PPA, or ACHA, and the infarct lesion on DWI conforms to one of the following characteristics (A, B, OR C):

A. LSA: "Comma-like" infarct lesions with "fan-shaped" extension from bottom to top in the coronary position OR ≥ 3 layers (layer thickness 5 mm) on axial DWI.

B. PPA: Infarct lesion extending from the deep pons to the ventral pons on axial DWI.

C. ACHA: Infarct within the anterior choroidal artery territory.

Exclusion Criteria:

* Typical recent small subcortical infarction (RSSI) (oval, <20mm in all axes)
* ≥ 50% stenosis on the parent artery (i.e., BA, MCA, or ICA)
* Stroke due to other clearly identified causes or possible cardioembolic etiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a BAD-related stroke, aged over 18 years, with symptom onset no more than 24 hours before admission, who were treated in one of the stroke units of the participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 462 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Favorable outcome (mRS 0-1) at three months. | Three months after acute ischemic stroke treatment
  Modified Rankin Scale (mRS) score at three months, with a favorable outcome defined as mRS 0-1 at three months.
Early neurological deterioration within 24-48 hours after symptom onset | within 24-48 hours after acute ischemic stroke onset
  Early neurological deterioration (END), defined as a worsening of the NIHSS score by ≥4 points within 24-48 hours after symptom onset.
Occurrence of symptomatic intracerebral hemorrhage. | within three months after acute ischemic stroke treatment.
  Occurrence of symptomatic intracerebral hemorrhage within three months after acute ischemic stroke treatment.

SECONDARY OUTCOMES:
Good functional outcome (mRS 0-2) | three months after acute ischemic stroke treatment.
  Modified Rankin Scale (mRS) score at three months, with a good outcome defined as mRS 0-2 at three months.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Frederic Hotz, DDr., Principal Investigator — 1. Department of Neurology, St. John's Hospital, Vienna, Austria, 2. Department of Neurology, University Hospital, Bern, Switzerland, 3. Department of Medicine I, Division of Infectious Diseases and Tropical Medicine, Medical University of Vienna, Vienna; Marek Sykora, Prof. Dr., Principal Investigator — 1. Sigmund Freud University Vienna, Austria, 2. Department of Neurology, St. John's Hospital, Vienna, Austria
Locations (7):
- Austria (2):
  - Department of Neurology, St. John's Hospital, Vienna, Austria, Vienna
  - Department of Neurology, Medical University of Vienna, Vienna
- Germany (3):
  - Department of Neurology, Berlin Institute of Health, Charité-Universitätsmedizin Berlin, Berlin
  - Department of Neurology, Heidelberg University Hospital, Heidelberg
  - Department of Neurology & Stroke, University of Tübingen, Tübingen
- Switzerland (2):
  - Department of Neurology, Universityhospital of Bern, Bern
  - Stroke Center, Neurology Service, Department of Clinical Neurosciences, Lausanne University Hospital and University of Lausanne, Lausanne

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification
Supporting Information: Study Protocol, SAP
Access Criteria: Data that support the findings of this study will available from the corresponding author after academic boards review and upon reasonable request

REFERENCES:
- [Background] Naimi AI, Whitcomb BW. Estimating Risk Ratios and Risk Differences Using Regression. Am J Epidemiol. 2020 Jun 1;189(6):508-510. doi: 10.1093/aje/kwaa044. No abstract available. PMID 32219364
- [Background] Barow E, Boutitie F, Cheng B, Cho TH, Ebinger M, Endres M, Fiebach JB, Fiehler J, Ford I, Galinovic I, Nickel A, Puig J, Roy P, Wouters A, Magnus T, Thijs V, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Simonsen CZ, Gerloff C, Thomalla G; WAKE-UP Investigators. Functional Outcome of Intravenous Thrombolysis in Patients With Lacunar Infarcts in the WAKE-UP Trial. JAMA Neurol. 2019 Jun 1;76(6):641-649. doi: 10.1001/jamaneurol.2019.0351. PMID 30907934
- [Background] Xu J, Xu X, Wang H, He L, Liu Q, Du Y, Wang J. Dual Antiplatelet Therapy Plus Argatroban Prevents Early Neurological Deterioration in Branch Atherosclerosis Disease. Stroke. 2022 Jan;53(1):e19-e20. doi: 10.1161/STROKEAHA.121.036356. Epub 2021 Nov 17. PMID 34784740
- [Background] Liu B, Zhang H, Wang R, Qu H, Sun Y, Zhang W, Zhang S. Early administration of tirofiban after urokinase-mediated intravenous thrombolysis reduces early neurological deterioration in patients with branch atheromatous disease. J Int Med Res. 2020 May;48(5):300060520926298. doi: 10.1177/0300060520926298. PMID 32459110
- [Background] Wu X, Liu Y, Nie C, Kang Z, Wang Q, Sun D, Li H, Liu Y, Mei B. Efficacy and Safety of Intravenous Thrombolysis on Acute Branch Atheromatous Disease: A Retrospective Case-Control Study. Front Neurol. 2020 Jul 7;11:581. doi: 10.3389/fneur.2020.00581. eCollection 2020. PMID 32733357
- [Background] Kobayashi Y, Kondo Y, Yamamoto K, Hirayama S, Kuasano Y, Tazawa KI, Shimizu Y, Sato A, Sekijima Y. Tissue plasminogen activator for acute branch atheromatous disease exhibits transient improvement and worsening. J Neurol Sci. 2024 Oct 15;465:123201. doi: 10.1016/j.jns.2024.123201. Epub 2024 Aug 30. PMID 39217764
- [Background] Yamamoto Y, Ohara T, Hamanaka M, Hosomi A, Tamura A, Akiguchi I. Characteristics of intracranial branch atheromatous disease and its association with progressive motor deficits. J Neurol Sci. 2011 May 15;304(1-2):78-82. doi: 10.1016/j.jns.2011.02.006. Epub 2011 Mar 13. PMID 21402390
- [Background] Duan Z, Fu C, Chen B, Xu G, Tao L, Tang T, Hou H, Fu X, Yang M, Liu Z, Zhang X. Lesion patterns of single small subcortical infarct and its association with early neurological deterioration. Neurol Sci. 2015 Oct;36(10):1851-7. doi: 10.1007/s10072-015-2267-1. Epub 2015 Jun 2. PMID 26032577
- [Background] Park MG, Oh EH, Kim BK, Park KP. Intravenous tissue plasminogen activator in acute branch atheromatous disease: Does it prevent early neurological deterioration? J Clin Neurosci. 2016 Nov;33:194-197. doi: 10.1016/j.jocn.2016.04.011. Epub 2016 Jul 21. PMID 27452127
- [Background] Nakase T, Yoshioka S, Sasaki M, Suzuki A. Clinical evaluation of lacunar infarction and branch atheromatous disease. J Stroke Cerebrovasc Dis. 2013 May;22(4):406-12. doi: 10.1016/j.jstrokecerebrovasdis.2011.10.005. Epub 2011 Nov 30. PMID 22133744
- [Background] Uchiyama S, Toyoda K, Kitagawa K, Okada Y, Ameriso S, Mundl H, Berkowitz S, Yamada T, Liu YY, Hart RG; NAVIGATE ESUS Investigators. Branch atheromatous disease diagnosed as embolic stroke of undetermined source: A sub-analysis of NAVIGATE ESUS. Int J Stroke. 2019 Dec;14(9):915-922. doi: 10.1177/1747493019852177. Epub 2019 May 27. PMID 31132967
- [Background] Adams HP Jr, Bendixen BH, Kappelle LJ, Biller J, Love BB, Gordon DL, Marsh EE 3rd. Classification of subtype of acute ischemic stroke. Definitions for use in a multicenter clinical trial. TOAST. Trial of Org 10172 in Acute Stroke Treatment. Stroke. 1993 Jan;24(1):35-41. doi: 10.1161/01.str.24.1.35. PMID 7678184
- [Background] Zhou L, Yao M, Peng B, Zhu Y, Ni J, Cui L. Atherosclerosis Might Be Responsible for Branch Artery Disease: Evidence From White Matter Hyperintensity Burden in Acute Isolated Pontine Infarction. Front Neurol. 2018 Oct 9;9:840. doi: 10.3389/fneur.2018.00840. eCollection 2018. PMID 30356780
- [Background] Kwan MW, Mak W, Cheung RT, Ho SL. Ischemic stroke related to intracranial branch atheromatous disease and comparison with large and small artery diseases. J Neurol Sci. 2011 Apr 15;303(1-2):80-4. doi: 10.1016/j.jns.2011.01.008. Epub 2011 Feb 1. PMID 21277587
- [Background] Petrone L, Nannoni S, Del Bene A, Palumbo V, Inzitari D. Branch Atheromatous Disease: A Clinically Meaningful, Yet Unproven Concept. Cerebrovasc Dis. 2016;41(1-2):87-95. doi: 10.1159/000442577. Epub 2015 Dec 16. PMID 26671513
- [Background] Caplan LR. Intracranial branch atheromatous disease: a neglected, understudied, and underused concept. Neurology. 1989 Sep;39(9):1246-50. doi: 10.1212/wnl.39.9.1246. No abstract available. PMID 2671793

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT07299994/Prot_SAP_000.pdf